CLINICAL TRIAL: NCT07046650
Title: Multi-cohort, Single-arm, Phase II Study of the Efficacy and Side Effects of Cisplatin Plus Gemcitabine in the Treatment of PD1 Failure or Intensive Treatment of Some Rare Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheng Zhang (Other)
Responsible Party: Sponsor-Investigator, Sheng Zhang, Dr., Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2501313
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rare Tumor 2 (Experimental): Patients with extramammary PAGET's disease, after PD1 failure.
  Interventions: Combination Product: cisplatin-based chemotherapy
- Rare Tumor 3 (Experimental): Patients with advanced adrenocortical carcinoma, following PD1 failure.
  Interventions: Combination Product: cisplatin-based chemotherapy
- Rare Tumor 4 (Experimental): Patients with advanced urachal cancer, after PD1 failure.
  Interventions: Combination Product: cisplatin-based chemotherapy
- Arm 1 (No Intervention): Patients with advanced urothelial cancer in whom PD-1 and vedicitumumab had failed.

INTERVENTIONS:
Combination Product: cisplatin-based chemotherapy — Patients were required to have a creatinine clearance of more than 60 and to receive standard doses of cisplatin and gemcitabine (gemcitabine 1000mg /m2 on day 1.8 and cisplatin 70 mg /m2 on day 1, q3w). A total of 4-6 courses of treatment were performed.
  Arms: Rare Tumor 2; Rare Tumor 3; Rare Tumor 4

SUMMARY:
This is a multi-cohort, single-arm, phase II study of the efficacy and side effects of cisplatin plus gemcitabine in the treatment of PD1 failure or intensive treatment of some rare tumors

DETAILED DESCRIPTION:
1. cisplatin plus gemcitabine regimen; Cisplatin-based chemotherapy, which is widely used in clinical oncology, is the cornerstone of many cancer treatments. Among them, it is extremely critical and important for germ cell tumors, especially testicular cancer, and for advanced urothelial cancer. In all treatment guidelines, cisplatin-based chemotherapy is used for advanced urothelial cancer. Cisplatin is also the most important drug in the treatment of testicular cancer, and it is an independent prognostic factor for the long-term survival of patients.

   The rapid development of immunotherapy, especially PD1, has made PD1 enter the front line of cancer treatment. It has become a first-line treatment typically for advanced urothelial cancer.

   "Advanced adrenocortical carcinoma, pheochromocytoma, extramammary PAGET's disease of the scrotum, advanced urachal carcinoma, and urinary sarcoma (after treatment with doxorubicin) are rare diseases for which standard treatment is lacking." However, PD1 is recommended by various guidelines due to its better safety.

   So, in the era of rapid changes in new treatment modalities, that is, after PD1 has entered the standard of care, does cisplatin-based chemotherapy still have corresponding anti-tumor activity?
2. treatment status of advanced bladder urothelial carcinoma Advanced bladder urothelial carcinoma (UC) is a highly fatal disease, and its treatment methods are diverse, but the effect is often limited by the metastatic site of the patient's tumor. In recent years, the rise of immunotherapy and ADC therapy has brought new hope to UC patients.

ADC drugs are a new direction in the field of urothelial cancer. A number of ADC drugs are available at home and abroad, including Enfortumab Vedotin (EV) 1, Sacituzumab Govitecan, and enfortumab vedotin. SG) and Disitamab Vedotin (RC48) have shown good efficacy in patients with advanced urothelial carcinoma after conventional treatment failure, and have become the treatment recommendation of guidelines and routine choice in clinical practice at home and abroad. ADC drug therapy may induce immunogenic cell death (ICD), thereby producing a synergistic anti-tumor effect with immunotherapy and further improving the efficacy. RC48 plus toripalimab: RC48-C014, a phase 1b/II study evaluating the efficacy and safety of RC48 plus toripalimab in patients with metastatic urothelial cancer, was updated at this meeting. A total of 32 patients were enrolled in the study, of which 28% had liver metastases, 62.5% had HER2 IHC(2+/3+), 37.5% had HER2 IHC(0/1+), and 56% had CPS≥1. In 20 patients with at least two responses, the confirmed ORR was 75% (95% CI, 50.9 to 91.3), with a CR rate of 15% and a DCR rate of 95% (95% CI, 75.1 to 99.9).

However, with the rapid change of treatment mode, the combination of ADC and PD1 has been confirmed in the EV3023,4 study, and the efficacy is much better than that of the traditional platinum-based first-line chemotherapy. This finding has led to a shift in the treatment of advanced urothelial carcinoai5 to first-line combination therapy with PD1 and EV, regardless of FDA approval or guidelines such as the NCCN.

In this context, first-line PD1 plus ADC therapy has become a game-changing new paradigm. However, the treatment of these patients after progression is still under controversy, and there is no relevant clinical research results to guide clinical practice.

A substantial number of patients in China choose these treatment modalities either as a result of enrollment in these clinical trials or on their own. A significant number of patients received first-line treatment with PD1 and ADC. However, since the active ingredient of vedicitumumab is anti-microtubule MMAE. Does the initial use of the drug affect the efficacy of subsequent platinum therapy? However, the toxicity of MMAE was mainly neurotoxicity. Platinum also has some neurotoxicity. So the toxicity effect on subsequent platinum therapy? Based on this, we designed the efficacy and safety of cisplatin combined with gemcitabine in patients with advanced urothelial carcinoma who had failed PD-1 and vedicitumumab treatment (arm 1). The efficacy of cisplatin plus gemcitabine was tested in individual rare cancers (arm II to arm IV).

2. Objectives of the study To determine the efficacy and safety of cisplatin combined with gemcitabine in some patients with pelvic tumors after standard treatment and PD1 failure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent was obtained before enrollment. 2. Age ≥18 years old; 3. Patients with corresponding cancer confirmed by histological and/or cytological examination; 4. Consent to treatment; 5. ECOG score: 0-1; 6. Previous PD-1 therapy failure; 7. At least one measurable lesion (≥10 mm on CT scan for non-nodal lesions and ≥15 mm on CT scan for nodal lesions according to RECIST criteria).

  8. Have adequate organ function: 9. Blood routine: Absolute Neutrophil Count (ANC) 1.5×109/L, Platelet (PLT) ≥70×109/L, Hemoglobin (HGB) ≥80g/L; 10. Liver function: serum Total Bilirubin (TBIL) ≤1.5× Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤3×ULN; Serum albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN; Patients who met the above criteria after conventional liver-protective therapy and could be stable for at least 1 week could be enrolled after investigator's evaluation.

  11. Renal function: creatinine clearance ≥60 mL/mi (using the standard Cockcroft-Gault formula) : 12. Coagulation: International Normalized Ratio (INR) ≤1.5 /PT≤1.5×ULN, aPTT≤1.5×ULN; If the subject is receiving anticoagulant therapy, as long as the PT and INR are within the prescribed range of anticoagulant drugs 13. Estimated survival time ≥3 months; 14. Contraception during treatment 15. Ability to adhere to study access schedules and other protocol requirements.

Exclusion Criteria:

* 1. Poor patient compliance; 2. Prior exposure to cisplatin and/or gemcitabine and documented progression 3. With ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (QTc≥470ms), and ≥ grade 2 congestive heart failure (New York Heart Association [NYHA] classification); 4. Severe active or uncontrolled infection (≥CTCAE grade 2 infection) requiring systemic antibacterial, antifungal, or antiviral therapy, including pulmonary tuberculosis infection.

  5. Active hepatitis (transaminase did not meet the inclusion criteria, hepatitis B reference: HBV DNA≥2000 IU/ml or ≥104 copies /ml; Hepatitis C reference: HCV RNA≥2000 IU/ml or ≥104 copies /ml; After nucleotide antiviral therapy, those below the above criteria can be enrolled). Chronic hepatitis B virus carriers with HBV DNA < 104 IU/ml could only be enrolled if they received antiviral therapy at the same time during the trial.

  6. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 7. Severe nausea, headache, insomnia, fatigue, somnolence, dry mouth, dizziness and constipation; 8. Patients with a history of active tuberculosis; 9. Patients who underwent major surgical treatment, open biopsy, or significant traumatic injury within 28 days before the initiation of study treatment; Or have a wound or fracture that has not healed for a long time; 10. Currently participating or having participated in another clinical investigator within 4 weeks before study initiation 11. Patients with a history of severe allergies 12. Is at risk for bleeding, or has coagulopathy, or is receiving thrombolytic therapy 13. People who have a history of psychotropic drug abuse and cannot quit or have mental disorders 14. Subjects who, in the investigator's judgment, had a concomitant medical condition that seriously compromised the safety of the subjects or interfered with the completion of the study, or who were deemed to be ineligible for enrollment for any other reason. "There was a clear previous history of neurological and psychiatric disorders, such as dementia, epilepsy, or seizure prone episodes.

  15. The presence of concomitant diseases (such as severe diabetes mellitus, thyroid disease, and psychosis), or serious and/or unstable medical, psychiatric, or other conditions (including laboratory abnormalities) that, in the judgment of the investigators, seriously compromise the safety of the subjects or prevent the subjects from completing the study, or the presence of serious and/or unstable medical, psychiatric, or other conditions (including laboratory abnormalities) that affect the safety of the patients or prevent the patients from providing informed consent, "Or the presence of any psychological, family, sociological, or geographic factors that affect the study protocol and follow-up plan.

  16. The investigator did not consider it appropriate to participate in the trial for any reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | through study completion, an average of 1 year
  The sum of the proportion of subjects with Complete response or Partial response

SECONDARY OUTCOMES:
Incidence of adverse events (AE) | through study completion, an average of 2 years
  Incidence of adverse events (AE)
During of response | through study completion, an average of 1 year
  The time between the start of the first assessment of the tumor as Complete response or Partial response and the second assessment as PD(Progressive Disease) or death from any cause
Progression Free Survival | through study completion, an average of 1 year
  The time, measured in days, from the date of first treatment to disease progression or death from any cause. Disease progression and death were measured in terms of preoccurrence. Progression included radiographic progression or clinical progression as assessed by the investigator.
Overall Survival | 2 years
  The time from the date of first treatment to death from any cause, measured in days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, Shanghai Municipality, China